CLINICAL TRIAL: NCT03659981
Title: Grey Matter Damage at the Earliest Phase of Multiple Sclerosis : a Longitudinal 7T Magnetic Resonance Imaging Study
Brief Title: Grey Matter Damage at the Earliest Phase of Multiple Sclerosis : a Longitudinal 7T MRI Study
Acronym: MSGM7T
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-01
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MS Patients (Experimental): Multiple sclerosis patients MRI 7T will be performed
  Interventions: Other: MRI 7T

INTERVENTIONS:
Other: MRI 7T — The imaging parameters will come from the 7 Tesla Siemens MRI

SUMMARY:
The present study is an opportunity to assess grey matter damage at the earliest phase of Multiple Sclerosis (MS) allowing to a better understanding of its origins and its impact and disease severity. This study is a preliminary longitudinal study to precisely depict the kinetic of grey matter damage and the links with disease aggravation. Thirty MS patients without time and spatial dissemination criteria (only one symptomatic MRI lesion detected) but with oligoclonal bands detected on cerebro spinal fluid analysis will be included for a monocentric transversal MRI study at 7T to assess grey matter injury. Clinical and neuropsychological assessments will be performed in the population the same day of a multi-parametric MRI. A longitudinal clinical and MRI follow up will be performed during 2 years.

DETAILED DESCRIPTION:
The present study is an opportunity to assess grey matter damage at the earliest phase of MS allowing to a better understanding of its origins and its impact and disease severity. This study is a preliminary longitudinal study to precisely depict the kinetic of grey matter damage and the links with disease aggravation. Thirty MS patients without time and spatial dissemination criteria (only one symptomatic MRI lesion detected) but with oligoclonal bands detected on cerebro spinal fluid analysis will be included for a monocentric transversal MRI study at 7T to assess grey matter injury. Clinical and neuropsychological assessments will be performed in the population the same day of a multi-parametric MRI. A longitudinal clinical and MRI follow up will be performed during 2 years.

ELIGIBILITY:
Inclusion Criteria:

* First presumed inflammatory demyelinating event in the central nervous system involving either the optic nerve, the spinal cord, a brain hemisphere, or the brainstem without spatial and time dissemination criteria
* Oligoclonal bands on CSF analysis
* Age between 18 and 45
* No previous history of neurological symptoms suggestive of demyelination
* No steroids in the month before MRI
* First MRI within six months after the first clinical episode

Exclusion Criteria:

* Possible alternative diagnoses
* Previous history of neurological or psychiatric disease
* Previous administration of immunosuppressive drugs
* Pregnancy
* Patient unable to give his consent for the study or patient under tutorship

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
number of cortical lesions | 2 hours
  Cortical lesion detection on 7T MRI at baseline

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France